CLINICAL TRIAL: NCT00474019
Title: A Phase I, Randomised, Open-label, Multi-National Study to Evaluate the Pharmacokinetics of Repeated Once-Daily Intravenous Doses of Esomeprazole in Paediatric Patients 0 to 17 Years Old, Inclusive.
Brief Title: Phase 1 Pharmacokinetics of Intravenous Nexium in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD, Nexium GI Established Brands, Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9615C00021
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Pharmacokinetics
Keywords: pediatrics; neonates
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Based on age and/or weight dose of esomeprazole IV qd in milligrams 20,40,10,20,10, 1.0 mg/kg, 0,5 mg/kg
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: esomeprazole — IV qd for 4 days
  Other Names: Nexium

SUMMARY:
The purpose of this research study is to evaluate how much of repeated once daily intravenous (IV, meaning through a vein) doses of esomeprazole gets into the bloodstream of hospitalized children aged 0-17 years old that require acid suppression therapy.

ELIGIBILITY:
Inclusion Criteria:

* parent/guardian must sign consent form and the child will be asked to sign and Assent Form if he/she is old enough and is able to sign
* verbal assent will be acceptable if the child is old enough to understand, but unable to write
* female and/or male hospitalized patients aged 0-17 years old who should be considered for treatment with acid suppressive therapy.

Exclusion Criteria:

* female patients that are pregnant, or plan to become pregnant during the study period or is breast-feeding a child
* patients with a history of multiple drug allergies
* any illness, medical history, abnormal laboratory values, abnormal physical examination findings or abnormal vitals signs that could put the patient at risk when participating in the study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2007-10; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic-area under plasma concentration versus time curve within a dosing interval | Day 4 of study

SECONDARY OUTCOMES:
Maximum plasma concentration, total, plasma clearance, steady-state volume of distribution of esomeprazole | Day 4 of study
Safety and tolerability will be assessed by AEs, laboratory values, blood pressure, heart rate, respiratory rate, body temperature, and ECG | Days 1-4 (during treatment), Days 1-28 (post treatment)
Evaluate main metabolites of esomeprazole (sulphone metabolite and 5-hydroxy metabolite) by assessment of max plasma conc, total area under the plasma concentration vs time curve within a dosing interval, clearance scaled by fraction metabolised | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Brown, MD, Study Director — AstraZeneca; Per Lundborg, MD, Study Director — AstraZeneca; Jill McGuinn, Study Director — AstraZeneca
Locations (15):
- United States (11):
  - Research Site, Little Rock, Arkansas
  - Research Site, Hartford, Connecticut
  - Research Site, Park Ridge, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Detroit, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, New Brunswick, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
- Research Site, North Adelaide, South Australia, Australia
- Research Site, Brussels (jette), Belgium, Belgium
- Research Site, Budapest, Hungary
- Research Site, Gothenburg, Sweden

REFERENCES:
- [Derived] Earp JC, Mehrotra N, Peters KE, Fiorentino RP, Griebel D, Lee SC, Mulberg A, Rohss K, Sandstrom M, Taylor A, Tornoe CW, Wynn EL, Van der Walt JS, Garnett C. Esomeprazole FDA Approval in Children With GERD: Exposure-Matching and Exposure-Response. J Pediatr Gastroenterol Nutr. 2017 Sep;65(3):272-277. doi: 10.1097/MPG.0000000000001467. PMID 27875488
- [Derived] Sandstrom M, Davidson G, Tolia V, Sullivan JE, Langstrom G, Lundborg P, Brown K. Phase I, multicenter, randomized, open-label study evaluating the pharmacokinetics and safety profile of repeated once-daily doses of intravenous esomeprazole in children 0 to 17 years of age. Clin Ther. 2012 Aug;34(8):1828-38. doi: 10.1016/j.clinthera.2012.06.028. Epub 2012 Jul 24. PMID 22832034